CLINICAL TRIAL: NCT00470288
Title: Randomized Controlled Trial of Bladder Flap vs.None
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mountain Area Health Organization Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-10-477
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-04

CONDITIONS: Cesarean Delivery Procedures
Keywords: cesarean delivery; bladder flaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bladder flap during cesarean section

SUMMARY:
Objective: To compare outcomes in cesarean section patients undergoing bladder flap versus none. Hypotheses: Operative time will be reduced with the elimination of a bladder flap during cesarean delivery and intra-operative and post-operative morbidity will not be significantly different.

Patients >= 35 wks gestation undergoing cesarean delivery will be randomized to bladder flap vs. none. Primary outcome is operative time (start to delivery); secondary outcomes include: injuries, EBL, intra-operative and post-operative complications,pain medication, hospital stay duration.

DETAILED DESCRIPTION:
1. Title A Randomized Controlled Trial of Bladder Flap vs. None in Cesarean Section
2. Background (This section should be used to provide a rationale for the conduct of the study. Refer to existent or preliminary studies as necessary) The standard of care in performing cesarean delivery is to perform a bladder flap in the procedures.1 The creation of a bladder flap essentially allows a surgeon to create a space between the uterus and the bladder so that he/she has better access to the lower portion of the uterus where a low transverse incision can be made. This procedure involves making a superficial incision into the peritoneum, or the cell lining of the abdominal cavity, and the moving the bladder down and away from the lower portion of the uterus. A retractor or a bladder blade is then inserted into this space to hold the bladder away from the uterus (see Appendix A).2 Use of the bladder flap in cesarean delivery dates back to 1878 in the pre-antibiotic era,3 and theoretically, the bladder flap allows better access to the low portion of the uterus while decreasing risk of bladder injury and infection. However, several recent but small studies suggest the inclusion of the bladder flap confers no advantage and may actually contribute to greater morbidity postoperatively. 4-5 Additionally, the incidence of bladder injuries is 0.3%, and most injuries resulted during the formation of the bladder flap.6 The evidence from these studies are limited by the inclusion of other modifications in surgical procedures and a lack of replication of results, respectively. Thus there is insufficient evidence to either support or reject the inclusion of bladder flaps in cesarean deliveries (Evidence grade C).7-8
3. Specific Objectives (Enumerate the objectives and nature of the measured end-points. Justify the use of surrogate clinical end-points as necessary)

1. To compare outcomes in cesarean section patients undergoing bladder flap versus none.

4. Study design (Explicate the nature of the study - observational vs experimental. Differentiate between cohort, case-control, and cross-sectional and randomized clinical trials. For the latter, provide sufficient supporting justification for the experimental arm. If it is a placebo-controlled trial, please state whether clinical equipoise exists between the placebo and experimental arm.) Randomized controlled trial.

Endpoints:

Total operating time (continuous) and Time of delivery to end of surgery (continuous) Estimated blood loss (continuous) Post operative fever (categorical) Bladder injury (categorical) Pre- and post-operative pain medication (continuous) and Analog pain scale (continuous)

5. Subject Selection (Include an enumeration of inclusion and exclusion criteria)

MAHEC patients presenting for delivery at Mission Hospitals requiring a cesarean section

Inclusion Exclusion Cesarean section All vaginal deliveries

≥ 35 weeks gestation < 35 weeks gestation Able to provide consent for medical treatment Urgent cesarean section Unable to provide consent for medical treatment Medical complications prohibitive of bladder flap Medical complications prohibitive of no bladder flap

6. Statistical methods, data analysis and interpretation (Include the factors considered in determining an appropriate sample size) Sample size of 100 per group based on an estimated mean difference of 5 minutes on total operating time (study arm 45±12.5 vs. bladder flap arm 50±12.5; Power=080; alpha=0.05; two-tailed).4

Per protocol analysis utilizing analysis of variance or for continuous variables and chi square analysis of categorical variables.

7. Study Procedures (Describe the chronological flow of the study, using schematic diagrams as necessary. Distinguish clearly between treatment-related [medically-indicated] and research-related procedures the subject will undergo)

All OB patients presenting at L&D for delivery will be approached for informed consent. consenting patients for whom a cesarean delivery is medically indicated will be randomized to bladder flap vs. none. Patients unable to consent for medical treatment or not wishing to consent for the project will be excluded. Consenting patients for whom a cesarean is medically indicated will be randomly assigned to bladder flap vs. by previously allocation of subject number. Patients will undergo assigned procedure unless excluded at the discretion of the surgeons who determine the alternate procedure is medically indicated. Patients undergoing the assigned procedure will have all data extracted from hospital medical records and entered into SPSS for a per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery at >=35 weeks gestation;
* Able to provide informed consent

Exclusion Criteria:

* Vaginal delivery;
* Delivery < 35 weeks gestation;
* STAT surgery;
* Unable to provide consent;
* Medical complication/condition incompatable with random asiignment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2005-10; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
operative time: start of surgery to delivery of infant | immediate: during cesarean surgery

SECONDARY OUTCOMES:
estimated blood loss | immediate
bladder injuries | immediate
other intra-operative complications | immediate
intra-operative transfusions | immediate
post-operative complications | post-op hospitalization
medication use: antibiotics and narcotics | post-op hospitalization
duration of post-op hospitalization | post-op hospitalization
readmisison post discharge | 6 weeks post-op

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Helms, MD, Principal Investigator — MAHEC OB/GYN; Shelley L Galvin, MA, Study Director — MAHEC OB/GYN
Locations (1):
- Mission Hospitals, Asheville, North Carolina, United States

REFERENCES:
- [Background] Hohlagschwandtner M, Ruecklinger E, Husslein P, Joura EA. Is the formation of a bladder flap at cesarean necessary? A randomized trial. Obstet Gynecol. 2001 Dec;98(6):1089-92. doi: 10.1016/s0029-7844(01)01570-8. PMID 11755558
- [Background] Wood RM, Simon H, Oz AU. Pelosi-type vs. traditional cesarean delivery. A prospective comparison. J Reprod Med. 1999 Sep;44(9):788-95. PMID 10509303
- [Background] Eisenkop SM, Richman R, Platt LD, Paul RH. Urinary tract injury during cesarean section. Obstet Gynecol. 1982 Nov;60(5):591-6. PMID 7145252